CLINICAL TRIAL: NCT00930176
Title: A Phase III Open, Multicentre Study to Investigate the Pharmacokinetics, Safety and Efficacy of BPL's High Purity Factor X in the Treatment of Severe and Moderate Factor X Deficiency.
Brief Title: A Study Investigating Treatment Factor X in People With Factor X Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ten01
Record Dates: First submitted 2009-06-10; First posted 2009-06-30 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Factor X Deficiency
MeSH Terms: conditions — Factor X Deficiency | interventions — Factor X

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human Coagulation FACTOR X (Experimental)
  Interventions: Biological: Human Coagulation FACTOR X

INTERVENTIONS:
Biological: Human Coagulation FACTOR X — Standard dose 25IU/kg to be administered at the Baseline Visit (1st PK assessment) and at the repeat PK assessment. Also administered to treat a bleed or to prevent a bleed.

SUMMARY:
The main objective of the study is to assess the pharmacokinetics of FACTOR X after a single dose of 25IU/kg.

The secondary objectives of the study are to assess efficacy and safety of FACTOR X in the treatment of bleeding episodes over at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given, or for subjects aged 12-17 years, have given written assent and whose parent/guardian has given written informed consent
* At least 12 years of age at dtae of written informed consent
* Have hereditary severe or moderate FX deficiency
* Currently treated with Fresh Frozen Plasma FFP, Prothrombin Complex Concentrate PCC or factor IX/X concentrate
* Must have a minimum of one spontaneous or menorrhagic bleed in the last 12 months which required treatment of FFP, PCC or factor IX/X concentrate. Newly diagnosed subjects who present at the hospital with a bleed may be included
* Must have had at least 7 days, and ideally 10-14 days, since an infusion of either FFP, PCC or factor IX/X concentrate at Baseline Visit
* Females of child bearing potential must have a negative result on a HCG based pregnancy test. If they are or become sexually active, they must practise contraception by using a method of proven reliability for the duration of the study

Exclusion Criteria:

* Have a history of inhibitor development to FX or a positive result at the Screening Visit
* Bleeding at the appointment for the PK assessment
* Subjects who have thrombocytopenia
* Have clinically significant liver disease
* Known to have other coagulopathy or thrombophilia
* Have known or suspected hypersensitivity to the investigational medicinal product or its excipients
* Have abused chemicals or drugs within the past 12 months
* Have a history of unreliability or non-cooperation
* Participating or have taken part in another trial within the last 30 days, with the exception of BPL FX surgery study - Protocol Ten03. In such cases, subjects should have completed their End of Study Visit either before or on the day of Screening Visit for this study
* Female subjects who are pregnant or lactating
* Subjects planning greater than 4 weeks absence from the locality of the Investigational site, between the screening visit and the repeat PK assessment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Shapiro, Dr, Principal Investigator — Co-Medical Director, Indiana Hemophilia and Thrombosis Center, 8402 Harcourt Road, Suite 420, Indianapolis, IN46260, USA
Locations (14):
- United States (3):
  - UCSF School of Medicine, San Francisco, California
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Dr. William Mitchell New York Blood Center, Weill Cornell Medical College, New York, New York
- Dr Gunter Auerswald, Bremen, Germany
- Spain (2):
  - Dr. Bermejo, Cáceres
  - Dr Maite Alvarez, Madrid
- Turkey (Türkiye) (6):
  - Cukurova University Hospital, Balcali, Adana
  - Ministry of Health Istanbul Goztepe Training & Research Hospital, Göztepe, Istanbul
  - Istanbul University Cerrahpasa School of Medicine, Istanbul
  - Kanuni Sultan Suleyman Training and Research Hospital, Istanbul
  - Prof. Kavakli, Izmir
  - Prof. Oner, Van
- United Kingdom (2):
  - Dr. Sue Pavord, Leicester
  - Dr. Steve Austin, London

REFERENCES:
- [Derived] Oner AF, Celkan T, Timur C, Norton M, Kavakli K. Use of a High-Purity Factor X Concentrate in Turkish Subjects with Hereditary Factor X Deficiency: Post Hoc Cohort Subanalysis of a Phase 3 Study. Turk J Haematol. 2018 May 25;35(2):129-133. doi: 10.4274/tjh.2017.0446. Epub 2018 Mar 16. PMID 29545231

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human Coagulation FACTOR X
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Human Coagulation FACTOR X
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 2
  Spain | 4
  Turkey | 6
  Germany | 1
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: FX:C Incremental Recovery
Description: Incremental recovery is defined as the peak rise in plasma FX levels (IU/dL), as measured at 15, 30 and 60 minutes post-dose, divided by the dose (IU/kg).
  Value given is the mean of 31 results: 16 for Baseline Visit + 15 for Repeat PK assessment
Time Frame: At Baseline (during first 60 minutes post-dose) and at 6 months post-Baseline (during first 60 minutes post-dose)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/dL per IU/kg
Arm/Group | Human Coagulation FACTOR X
Number analyzed (Participants) | 16
IU/dL per IU/kg | 2.07 (21.01)

2. Primary Outcome: FX:C Half-life
Description: Value given is the mean of 31 results: 16 for Baseline Visit + 15 for Repeat PK assessment
Time Frame: At Baseline and at 6 months post-Baseline
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Human Coagulation FACTOR X
Number analyzed (Participants) | 16
hours | 29.36 (22.89)

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 28 days post-last dose.
Arm/Group | Human Coagulation FACTOR X
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Coagulation FACTOR X (N=16)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastric ulcer helicobacter (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Coagulation FACTOR X (N=16)
Haematoma (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 4 (4)
Urticaria (Immune system disorders) | 1 (2)
Fatigue (General disorders) | 1 (2)
Infusion site erytema (General disorders) | 1 (2)
Infusion site pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (2)
Swelling (General disorders) | 1 (1)
Ulcer (General disorders) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (14)
Migraine (Nervous system disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6)
Odynophagia (Gastrointestinal disorders) | 1 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (11)
Oral infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (9)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days